CLINICAL TRIAL: NCT03078270
Title: A Controlled Study of the Efficacy of Botulinum Toxin A (Botox) for the Treatment of Social Anxiety Disorder (SAD)
Brief Title: A Study of the Efficacy of Botox in the Treatment of Social Anxiety Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: study terminated due to low recruitment
Sponsor: Daniel Lieberman (Other)
Responsible Party: Sponsor-Investigator, Daniel Lieberman, Physician Faculty Director, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 041641
Record Dates: First submitted 2017-02-21; First posted 2017-03-13 (Actual); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Anxiety Disorder Social; Anxiety
Keywords: social anxiety; botulinum toxin; botox
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Open-label (Other): 10 participants will be recruited for an open-label study. All will receive the active medication and complete depression and anxiety surveys at baseline, 4-weeks, and 8-weeks post injection. All participants will receive botulinum toxin A.
  Interventions: Drug: botulinum toxin A
- Double-Blind (Placebo Comparator): 30 participants will be recruited for a double-blind, comparison study. Participants will be randomized to the active or control groups. Each will receive an injection (active medication or placebo) and will complete a depression and anxiety survey at baseline, 4-weeks and 8-weeks post injection. Participants in the active group will receive botulinum toxin A; participants in the control group will receive a placebo.
  Interventions: Drug: botulinum toxin A; Other: Placebo

INTERVENTIONS:
Drug: botulinum toxin A — Single treatment visit for 5 injections of botulinum toxin A, 40 units (for females) and 50 units (for males)/
  Other Names: Botox
Other: Placebo — single treatment visit for 5 injections of normal saline
  Other Names: Saline
  Arms: Double-Blind

SUMMARY:
The goal of this study is to see whether Botox is an effective treatment for social anxiety disorder (SAD). Participants will complete two short surveys on depression and anxiety symptoms, receive a one-time injection of Botox, and complete the depression and anxiety survey 4 weeks after injection and again at 8 weeks after injection.

DETAILED DESCRIPTION:
The use of botulinum toxin A to correct glabellar frown lines is an effective and popular cosmetic procedure with more than 1 million treatments per year in the United States alone (Carruthers, A.). Botulinum toxin type A marketed commercially as BOTOX® Cosmetic (Botox), is produced from fermentation of Hall strain Clostridium botulinum type A grown in a medium containing casein hydrolysate, glucose, and yeast extract, intended for intramuscular use.

Botox blocks neuromuscular transmission by binding to acceptor sites on motor nerve terminals, entering the nerve terminals, and inhibiting the release of acetylcholine. When injected intramuscularly at therapeutic doses, Botox produces partial chemical denervation of the muscle resulting in a localized reduction in muscle activity. In addition, the muscle may atrophy, axonal sprouting may occur, and extrajunctional acetylcholine receptors may develop. There is evidence that reinnervation of the muscle may occur, thus slowly reversing muscle denervation produced by Botox.

Botox is indicated for the temporary improvement in the appearance of moderate to severe glabellar lines associated with corrugator and/or procerus muscle activity in adult patients ≤ 65 years of age.

Botox is contraindicated in the presence of infection at the proposed injection site(s) and in individuals with known hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation.

Depression

The first open label trial of Botox to the glabellar muscle complex to treat unipolar depression was published in 2006. Since that time, three randomized double blind placebo-controlled trials were conducted to assess the efficacy of Botox treatment of the glabellar muscle complex in major depression. All three studies showed a response rate of 50 to 60%, and the remission rate of approximately one-third. To date, no clinical trials of Botox have been conducted in SAD.

Social Anxiety Disorder (SAD)

Social anxiety disorder (SAD) is a common psychiatric condition marked by persistent fear and anxiety of one or more social or performance situations. The lifetime prevalence of the disorder is 12%, and leads to significant morbidity for those affected. The only FDA approved treatments for SAD have response rates of 40 to 60 %, and remission rates of 20%. Therefore, there is a real need for the development of new and effective treatments for SAD.

Patients suffering from SAD either avoid situational triggers or endure intense anxiety and distress, leading to an impaired social life in either scenario. SAD is characterized by an overactive anxiety pathway with a perceptual and cognitive bias towards threat.

The amygdala, a limbic region with multiple projections to cortical and subcortical regions, is thought to be critically involved in the regulation of emotion, with a general role in directing attention to affectively salient stimuli, recruiting and coordinating cortical arousal for optimizing sensory and perceptual processing of ambiguous or novel stimuli.. A tight link between fear and the amygdala has been suggested. Fear related neuronal circuits involving the amygdala are thought to play a role in the generation of social withdrawal, fear, and anxiety.

Recently, two studies have linked botulinum toxin A treatment of the frown with down-regulation of amygdala activity. Patients who received botulinum toxin A injections into their frown muscles had decreased activity in the amygdala and its coupling with brain stem activity when mimicking angry facial expressions. Further research has confirmed that amygdala activity in response to angry faces was decreased when the frown muscles were paralyzed by botulinum toxin A injection. Furthermore, amygdala activity returned to its original state after the effects of the botulinum toxin A injection had worn off, confirming that botulinum toxin A reversibly severed afferent feedback from the corrugator muscle to the amygdala.

Given that SAD patients show abnormal patterns of amygdalar activation after viewing emotional faces, we believe that there is a good likelihood that some of the symptoms of SAD will improve after botulinum toxin A treatment of the frown.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of social anxiety disorder
* women of childbearing potential on an acceptable form of birth control and are not pregnant or lactating

Exclusion Criteria:

* has ever been treated with botulinum toxin A
* has another Axis I diagnosis within in the 6-months prior to screening
* history of substance abuse within 2-months of screening
* current or recent suicidality
* scoring greater than 2 on Beck Depression Inventory (BDI) suicidality question
* psychotic or bipolar disorder
* unstable medical condition
* changes in medication or psychotherapy treatment in the month prior to screening
* significant risk of committing homicide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Z Lieberman, MD, Principal Investigator — George Washington University
Locations (1):
- GW University Medical Faculty Associated, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing is not planned on being shared with other investigators

REFERENCES:
- [Background] Reichenberg JS, Hauptman AJ, Robertson HT, Finzi E, Kruger TH, Wollmer MA, Magid M. Botulinum toxin for depression: Does patient appearance matter? J Am Acad Dermatol. 2016 Jan;74(1):171-173.e1. doi: 10.1016/j.jaad.2015.08.051. No abstract available. PMID 26702796
- [Background] Finzi E, Wasserman E. Treatment of depression with botulinum toxin A: a case series. Dermatol Surg. 2006 May;32(5):645-9; discussion 649-50. doi: 10.1111/j.1524-4725.2006.32136.x. PMID 16706759
- [Background] Finzi E, Rosenthal NE. Emotional proprioception: Treatment of depression with afferent facial feedback. J Psychiatr Res. 2016 Sep;80:93-96. doi: 10.1016/j.jpsychires.2016.06.009. Epub 2016 Jun 16. PMID 27344227
- [Background] Magid M, Reichenberg JS, Poth PE, Robertson HT, LaViolette AK, Kruger TH, Wollmer MA. Treatment of major depressive disorder using botulinum toxin A: a 24-week randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2014 Aug;75(8):837-44. doi: 10.4088/JCP.13m08845. PMID 24910934
- [Background] Wollmer MA, de Boer C, Kalak N, Beck J, Gotz T, Schmidt T, Hodzic M, Bayer U, Kollmann T, Kollewe K, Sonmez D, Duntsch K, Haug MD, Schedlowski M, Hatzinger M, Dressler D, Brand S, Holsboer-Trachsler E, Kruger TH. Facing depression with botulinum toxin: a randomized controlled trial. J Psychiatr Res. 2012 May;46(5):574-81. doi: 10.1016/j.jpsychires.2012.01.027. Epub 2012 Feb 24. PMID 22364892

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label: 4 participants were recruited for the open-label study.
- Double-Blind: 0 participants were recruited for the double-blind, comparison study.
Period: Overall Study
Arm/Group | Open-label | Double-Blind
Started | 4 | 0
Completed | 0 | 0
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Population: No participants were recruited into the double blind study
Groups:
- Open-label: 4 participants were recruited with social anxiety disorder.
- Double-Blind: No participants were recruited.
- Total: Total of all reporting groups
Arm/Group | Open-label | Double-Blind | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants] — 18-65
  Participants
    <=18 years | 0 |  | 0
    Between 18 and 65 years | 4 |  | 4
    >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of of Botulinum Toxin A Reducing Symptoms of Social Anxiety Disorder
Description: Repeated measure at baseline, 4-weeks and 8-weeks post-injection of anxiety using the Liebowitz Social Anxiety Scale to determine treatment response.
Time Frame: 2 months
Population: The study was closed before outcome measures were collected.
Arm/Group | Open-label | Double-Blind
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 11 months
Description: No adverse events were reported.
Arm/Group | Open-label | Double-Blind
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT03078270/Prot_SAP_000.pdf